CLINICAL TRIAL: NCT04108975
Title: Assessment of the Effect of Rectus Muscle Reapproximation Versus Non Reapproximation During CS on Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelraheem Ali, Obstetrician, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Rectus muscle reapproximation
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectus muscle reapproximation group (Active Comparator): Rectus muscle reapproximation by 3 interrupted simple sutures or 3 vertical mattress sutures
  Interventions: Procedure: Rectus muscle reapproximation during CS
- Rectus muscle non reapproximation group (Active Comparator): No rectus muscle reapproximation will be done based on the fact that rectus muscle can regain its position
  Interventions: Procedure: Rectus muscle non reapproximation during CS

INTERVENTIONS:
Procedure: Rectus muscle reapproximation during CS — Reapproximation by 3 interrupted simple sutures or 3 vertical mattress sutures.
  Arms: Rectus muscle reapproximation group
Procedure: Rectus muscle non reapproximation during CS — During CS rectus muscle non reapproximation will be done.
  Arms: Rectus muscle non reapproximation group

SUMMARY:
The aim of this study is to assess the effect of rectus muscle re-approximation by 3 interrupted simple sutures versus tighting it by 3 vertical mattress sutures during cesarean delivery on postoperative pain.

DETAILED DESCRIPTION:
In recent years, Cesarean deliveries have increased dramatically worldwide. In Egypt, 52% of women give birth by Cesarean Section according to the 2014 Demographic and Health survey. Despite the rising incidence of Cesarean section, controversy about the optimal surgical method of Cesarean section still remains. Obstetricians use a variety of surgical techniques to reduce post-operative adhesions after Cesarean section, such as parietal peritoneal closure and rectal muscle approximation. They believe that adhesions may result from exposure of an opened intraperitoneal cavity to the subfascial space which can be prevented by approximating the rectus muscle or closing the parietal peritoneum. In addition, rectus muscle approximation may be considered to reduce the risk of persistent rectus muscle diastasis. However, different studies showed a controversy and inconsistency in the practice of rectus muscle re-approximation among surgeons. Some obstetricians agree that the rectus muscles can regain their right anatomic position by themselves and that suturing them together does not add any benefit. Even though, one of their main concern against rectus muscle approximation is its potential association with increased post operative pain, hence the importance of this prospective randomized controlled study. The aim of the investigator's study is to assess the effect of rectus muscle re-approximation by 3 interrupted simple sutures versus tighting it by 3 vertical mattress sutures during cesarean delivery on postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* • Primigravida

  * Single pregnancy
  * Term at >37 weeks
  * Maternal age between 18 and 35 yrs
  * Spinal anaesthesia.
  * No other medical diseases.

Exclusion Criteria:

* • prior laparotomy

  * vertical skin incision
  * chronic analgesia use
  * allergy to opioid or nonsteroidal anti-inflammatory drugs
  * body mass index more than or equal to 40.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 156 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain: 4 point verbal rating scale (VRS) | 1 week after operation
  Post-operative pain is analyzed by using 4 point verbal rating scale (VRS) which consists of a list of adjectives describing different levels of pain intensity i.e (no pain =1, mild pain = 2, moderate pain = 3, severe pain = 4), patients are asked to read this list of adjectives and select the word that best describes their level of pain on the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Aboalfadl, Professor, Study Director — Assiut University; Diaa Abdelaal, Professor, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No